CLINICAL TRIAL: NCT05236582
Title: Herombopag for Chemotherapy-induced Thrombocytopenia: a Prospective Multi-center One-arm Study in Solid Tumors
Brief Title: Herombopag for Chemotherapy-induced Thrombocytopenia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Tianjin Medical University Cancer Institute and Hospital (Other); Tianjin Medical University Second Hospital (Other); Tianjin Third Central Hospital (Other); Tianjin People's Hospital (Other); Henan Cancer Hospital (Other Government); The Second Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2020014（Herombopag）
Record Dates: First submitted 2022-01-20; First posted 2022-02-11 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Chemotherapy-induced Thrombocytopenia; Herombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 50 subjects with chemotherapy-induced thrombocytopenia (Experimental): 50 enrolled subjects will be picked up to take Herombopag at the indicated dose.
  Interventions: Drug: Herombopag

INTERVENTIONS:
Drug: Herombopag — The subjects will initiate treatment with 7.5 mg/d Herombopag. Platelet counts is obtained weekly and dose adjustment should be done according to platelet counts, and maximum dose should not exceed 7.5 mg daily. Subjects whose platelet count ≤100×109/L，the Herombopag dose will maintain. If platelet count >100×109/L for 2 weeks, the subjects need to reduce the dose of Herombopag to the next lower dose or lower frequency. If subjects whose platelet count exceeds 100×109/L for 4 weeks，already have reduced the dose of Herombopag to 2.5mg once every other day or lower frequency during the treatment period, Herombopag can be stopped for observation, until platelet counts fall below 100×109/L. If the subjects do not need further chemotherapy or radiotherapy, the subjects can taper off Herombopag if the platelet is greater than 50×109/L.

SUMMARY:
To evaluate the efficacy and safety of Herombopag to treat chemotherapy-induced thrombocytopenia in Solid Tumors

DETAILED DESCRIPTION:
The investigator had registered a clinical trial of Eltrombopag in the treatment of chemotherapy-induced thrombocytopenia（NCT04600960）. Due to the late launch of Herombopag in China, the investigator also collected the information of Herombopag in the treatment of chemotherapy-induced thrombocytopenia according to the protocal of Eltrombopag in the treatment of chemotherapy-induced thrombocytopenia（NCT04600960）.

This is a single-arm study to evaluate the safety and efficacy of Herombopag to treat chemotherapy-induced thrombocytopenia（CIT）. These subjects have been treated with recombinant human thrombopoietin（rhTPO） or interleukin 11（IL-11） before, the platelets can rise to normal or reach the effective standard, but after the re-application, the effective standard is not reached, or the effective standard is still not reached after the rhTPO 300U/kg/d treatment for 14 days. The investigator will assess the changes of the platelet counts after the treatment of Herombopag from week 1 to week 24, and observe incidence of adverse events during the treatment of Herombopag. The investigator will complete the 4 weeks safety visits（once a week），if the subjects end or withdraw from the clinical trial.

Patients with chemotherapy-induced thrombocytopenia who had the same inclusion and exclusion criteria in the same period or in the past will be compared with the efficacy and safety of supportive treatment and Eltrombopag or Avatrombopag treatment in the same period or history, so as to preliminarily explore and evaluate the efficacy and safety of Herombopag treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years old, male or female;
* Conform to the diagnostic criteria of chemotherapy-induced thrombocytopenia (CIT); Ineffective after repeated treatment with rhTPO or IL-11；
* Stop radiotherapy or chemotherapy for more than 1 month;
* Platelet counts <30 ×10^9/L, and bleeding tendency;
* Estimated survival period ≥ 6 months；
* People who are willing to sign the informed consent voluntarily and follow the research program.
* Liver and kidney function<1.5×upper limit of normal, qualified for physical examination；
* Subject is practicing an acceptable method of contraception. Women of childbearing potential must have a negative serum pregnancy test in the whole study;

Exclusion Criteria:

* Those with uncontrollable primary diseases of important organs, such as extensive metastasis of malignant tumors, liver failure, heart failure, kidney failure and other diseases；
* Patients with poor compliance;
* Positive serology for HIV, hepatitis B virus (HBV), hepatitis C virus (HCV), and/or hepatitis D virus (HDV), Syphilis; Positive for Epstein-Barr Virus DNA, Cytomegalovirus DNA;
* Accompanied by extensive and severe bleeding, such as hemoptysis, upper gastrointestinal bleeding, intracranial hemorrhage, etc.
* There is currently a heart disease requiring treatment or a poorly controlled hypertension judged by the investigator；
* Patients with thrombotic diseases such as pulmonary embolism, thrombosis, and atherosclerosis；
* Those who have received allogeneic stem cell transplantation or organ transplantation in the past；
* Patients with mental disorders who cannot normally obtain informed consent and undergo trials and follow-up；
* Patients whose toxic symptoms caused by treatment before participating in the trial have not disappeared；
* Other serious diseases that may restrict participants from participating in this trial (such as diabetes; severe heart failure; myocardial obstruction or unstable arrhythmia or unstable angina in the past 6 months; gastric ulcers; mobility Autoimmune diseases, etc.)；
* Patients with sepsis or patients with other irregular bleeding；
* Patients taking antiplatelet drugs at the same time；
* Pregnant women, suspected pregnancy (a positive pregnancy test for human chorionic gonadotropin in urine at screening) and breastfeeding patients；
* Pre-existing cardiac disease, including congestive heart failure of New York Heart Association [NYHA] Grade III/IV, arrhythmia requiring treatment or myocardial infarction within the last 6 months. No arrhythmia known to increase the risk of thrombotic events (e.g. atrial fibrillation), or patients with a QT >450msec or QTc > 480 for patients with a Bundle Branch Block;
* Researchers believe that patients should not participate in the test of any other condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of the platelet counts after the treatment of Herombopag at week 12 | 12 weeks
  The investigator will assess the changes of the platelet counts after the treatment of Herombopag from week 1 to week 24，and calculate the proportion of subjects ≥ 30 × 10^9/L ， 50 × 10^9/L and 100 × 10^9/L at week 12.
Changes of the platelet counts after the treatment of Herombopag at week 24 | 24 weeks
  The investigator will assess the changes of the platelet counts after the treatment of Herombopag from week 1 to week 24，and calculate the proportion of subjects ≥ 30 × 10^9/L ， 50 × 10^9/L and 100 × 10^9/L at week 24.

SECONDARY OUTCOMES:
Incidence of adverse events after the treatment of Herombopag | 24 weeks
  The investigator will observe incidence of adverse events after the treatment of Herombopag, including thrombosis, diarrhea, skin rash, abnormal liver function and so on.
Changes of concentration of TPO in peripheral blood | 24 weeks
  The investigator will observe the concentration of TPO in peripheral blood before and after the treatment of Herombopag, if necessary.
Changes of concentration of TPO antibodies，anti-c-Mpl antibodies and TPO neutralizing antibodies in peripheral blood | 24 weeks
  The investigator will observe the concentration of antibodies in peripheral blood before and after the treatment of Herombopag, if necessary

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Principal Investigator — Chinese Academy of Medical Science and Blood Disease Hospital
Locations (1):
- Chinese Academy of Medical Science and Blood Disease Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Researchers qualified can request the dataset, including de-identified individual subject data. Data may be requested from PI from 12 months 36 months after study completion.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months to 36 months after study completion.
Access Criteria: Upon request to PI.